CLINICAL TRIAL: NCT06236386
Title: Translating Virtual Reality Research Evidence Into Clinical Practice During Colonoscopy Procedures
Brief Title: Virtual Reality During Colonoscopy Procedures
Acronym: VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Sherily Pereira-Morales, Principal Investigator, University of Puerto Rico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-05-102
Record Dates: First submitted 2023-10-04; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a convergent mixed methods (QUAN + QUAL) design to measure the reach, effectiveness, adoption, implementation, and maintenance of translating VR evidence into practice.
  Qualitative data will be collected after the colonoscopy procedure by using a customized satisfaction survey, measuring the experience and satisfaction of patients and clinicians. Six months after launching this study, clinicians will be surveyed about their continuation of using VR during colonoscopy procedures.
  Individual quantitative and qualitative results will be merged initially through a convergent data analysis integration strategy that will compare both strands side by side. This strategy contributes to the overall interpretation of the findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Experience (Other): A VR headset will be loaned to patients to be immersed in a VR environment while undergoing their colonoscopy.
  Interventions: Other: VR Experience

INTERVENTIONS:
Other: VR Experience — VR headset and video experience.

SUMMARY:
Colorectal cancer (CRC) in the United States (US) is the fourth leading cause of cancer- related deaths. In Puerto Rico (PR), the incidence and mortality rate of CRC is higher (41% and 14%) in comparison to the mainland US (38% and 13%). To reduce mortality, receiving a colonoscopy is considered the gold standard for early detection. Yet Puerto Ricans are less likely to adhere to this recommendation than individuals in the mainland US (52% vs. 65%).

Fear of acute pain may contribute to this reluctance despite the administration of sedation and analgesia during the procedure. The American Society for Gastrointestinal Endoscopy's recommended current standard of practice is to administer opioids and benzodiazepines to achieve minimal and/or moderate sedation during a colonoscopy procedure. Because patients still have conscious awareness, adding an effective pain distraction tool, such a virtual reality (VR), to their pharmacological standard of care during this short procedure could improve outcomes through decreased opioid and anxiolytic administration.

Strong evidence supports VR's effectiveness to distract patients from acute pain during brief medical procedures. To address this translational gap from research to clinical practice within a Hispanic oncology population receiving colonoscopies, an implementation science (IS) framework will be utilized to measure: reach, effectiveness, adoption, implementation, and maintenance. RE-AIM is an IS framework that systematically measures and supports sustainable adoption and implementation of evidence-based interventions into clinical practice. The purpose of this IS study will be to evaluate the translation of VR into clinical practice for patients during a CRC screening colonoscopy.

DETAILED DESCRIPTION:
The purpose of this study will be to evaluate the translation of VR into clinical practice for patients scheduled to receive a CRC screening through a colonoscopy. Findings from this study has widespread implications of translating VR technology to other patient populations and clinical settings during short procedures to improve outcomes. The specific aims will be to:

Aim 1. Determine the feasibility of implementing a VR distraction experience for patients during colonoscopy procedures using the RE-AlM framework. Using a mixed-methods approach, the investigators will evaluate participant participation (reach), opioid and benzodiazepines use, pain and sedation scores before, during, and after the procedure (effectiveness), acceptance of the VR experience (adoption), use of VR experience as intended (implementation), and continued long-term use of VR (maintenance) through quantitative and qualitative measurements.

Aim 2. Determine the costs and return on investment of implementing a VR experience for patients during colonoscopy procedures. The investigators will evaluate and compare the cost of the VR intervention and the rate of adverse events related to opioid administration to calculate return on investment.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive a colonoscopy procedure
* 21 years of age or older
* Ability to read and speak in Spanish.

Exclusion Criteria:

* History of seizures
* Balance disorder
* Current infectious disease
* Cognitive and visual impairments
* Sedation intolerance
* History of motion sickness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Level of Pain | 10 months
  Numeric Rating Scale: 0 (No Pain) to 10 (worst possible pain)
Ramsay Score | 10 months
  Ramsay score: 1 to 6 (1- Awake; agitated or restless or both to 6-sleep; Asleep; no response to glabellar tap or loud auditory stimulus)
Medication Administration | 10 months
  Medications administered: opioids, benzodiazepines, other medication
Procedure Length | 10 months
  Length of the procedure: minutes
Recovery Time | 10 months
  Recovery time: minutes
Preferred Video Type | 10 months
  VR video type: video content (ocean, nature, space)
VR Experience satisfaction | 10 months
  VR Experience satisfaction questions: 5-point Likert scale (1-Strongly disagree - 5 Strongly agree)
Clinician Feedback | 10 months
  Clinician Open-ended question about what would be changed from the process

SECONDARY OUTCOMES:
Length of recovery | 10 months
  Length of time in Recovery (minutes)
Adverse Events | 10 months
  Frequency of adverse events (name and number)
Medication Use | 10 months
  Medication administration comparison between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sherily Pereira, PhD, FAAN, Principal Investigator — University of Puerto Rico, Medical Sciences Campus, School of Nursing

IPD SHARING:
Plan to Share IPD: No